CLINICAL TRIAL: NCT01699178
Title: Open-Label Study of Oral Testosterone Undecanoate (TU) in Hypogonadal Men
Brief Title: Open-label, Follow-up Study of Oral Testosterone Undecanoate in Hypogonadal Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAR-12010
Record Dates: First submitted 2012-09-05; First posted 2012-10-03 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Male Hypogonadism
MeSH Terms: conditions — Eunuchism | interventions — testosterone undecanoate; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral testosterone undecanoate (Experimental): Oral testosterone undecanoate; continue dose from previous Phase III trial; 100-300 mg T (as TU), BID, for 12 months.
  Interventions: Drug: Oral testosterone undecanoate
- Transdermal testosterone gel (AndroGel) (Active Comparator): Transdermal testosterone gel; continue dose from previous Phase III trial, 2.5-10 g/applied once daily for 12 months
  Interventions: Drug: Transdermal testosterone gel (AndroGel)

INTERVENTIONS:
Drug: Oral testosterone undecanoate — Total daily dose of T = 200 mg T (as 316 mg TU) to 600 mg T (as 948 mg TU), taken as 100 mg to 300 mg T BID
  Other Names: Oral TU
  Arms: Oral testosterone undecanoate
Drug: Transdermal testosterone gel (AndroGel) — Total daily dose of T = 2.5 to 10 g of gel (25 mg to 100 mg T) QD
  Other Names: AndroGel
  Arms: Transdermal testosterone gel (AndroGel)

SUMMARY:
The purpose of this one year extension (follow-up) study is to gather additional safety data in hypogonadal men treated with oral TU or AndroGel who have completed the 12-month Phase III study CLAR-09007.

DETAILED DESCRIPTION:
This is the long-term extension of Study CLAR-09007, which like Study CLAR-09007, is an open-label study. This study contained an arm to evaluate the oral TU formulation as well as a comparator arm of the market-leading transdermal T-gel formulation. The comparator arm was included in the Phase III study and in this extension study to allow a general evaluation of comparative safety. Subjects randomized to oral TU in the Phase III study were continued on oral TU in the extension, and those who completed this 12-month Phase IV study have been followed for a total of 2 years of oral TU therapy. Likewise, subjects randomized to transdermal T-gel in the Phase III study were continued on T-gel in the extension, and those who completed this 12-month Phase IV study have been followed for a total of 2 years of T gel therapy. This 2-year period of therapy and assessments was to provide a long-term view of the safety of oral TU and the stability of the T replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects were to have completed Study CLAR-09007.
2. Subjects were to have adequate venous access in the left or right arm to allow collection of a number of blood samples via a venous cannula.
3. Subjects were required to remain off all forms of T except for study medication throughout the entire study.
4. Subjects voluntarily gave written informed consent to participate in this study.

Subjects meeting any of the following criteria were not eligible for participation in this study:

1. Significant intercurrent disease of any type, in particular liver, kidney, uncontrolled or poorly controlled heart disease, or psychiatric illness developed during the Phase III study that would, in the opinion of the Investigator, require exclusion from this study.
2. Untreated, severe obstructive sleep apnea (diagnosed during previous Phase III study).
3. Serum transaminases >2 times upper limit of normal (ULN), serum bilirubin >2.0 mg/dL and serum creatinine >2.0 mg/dL at the final visit for Study CLAR 09007.
4. Abnormal prostate digital rectal examination (palpable nodule[s]) or elevated PSA (serum PSA >4 ng/mL) at the final visit for Study CLAR-09007.
5. Use of dietary supplement saw palmetto or phytoestrogens and use of any dietary supplements that may increase serum T, such as androstenedione or dehydroepiandrosterone (DHEA).
6. Known malabsorption syndrome and/or current treatment with oral lipase inhibitors (e.g., orlistat [Xenical]) and bile acid-binding resins (e.g., cholestyramine [Questran], colestipol [Colestid]).
7. Poor compliers with study medication, study procedures, or study visits in Study CLAR 09007.
8. Concomitant use of antiandrogens, estrogens, potent oral CYP3A4 inducers (e.g., barbiturates, glucocorticoids [pharmacologic doses of glucocorticoids for replacement therapy were not exclusionary]) and potent CYP3A4 inhibitors (e.g., human immunodeficiency virus [HIV] antivirals [indinavir, nelfinavir, ritonavir, saquinavir, delaviridine], amiodarone, azithromycin, ciprofloxacin, ketoconazole). (Note: Short-term ciprofloxacin administration completed more than 7 days prior to study visits was not exclusionary during the study.)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Swerdloff, MD, Principal Investigator — University of California, Los Angeles
Locations (30):
- United States (25):
  - Alabama Clinical Therapeutics, Inc., Birmingham, Alabama
  - Alabama Internal Medicine, PC, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Calera, Alabama
  - Medical Affiliated Research Center, Inc, Huntsville, Alabama
  - Quality of Life Medical and Research Centers, LLC, Tucson, Arizona
  - Providence Clinical Research, Burbank, California
  - South Orange County Endocrinology, Laguna Hills, California
  - Tower Urology, Los Angeles, California
  - David Geffen School of Medicine, UCLA, Los Angeles, California
  - Harbor-UCLA Medical Center, LA Biomedical Research Institute, Torrance, California
  - Connecticut Clinical Research Center/ConnecTrials, Middlebury, Connecticut
  - University of CT School of Medicine, New Haven, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Maimonides Medical Center, Brooklyn, New York
  - Bruce R. Gilbert, MD, PhD, Great Neck, New York
  - University Urology Associates, New York, New York
  - Michael A. Werner, Purchase, New York
  - Sunstone Medical Research, Medford, Oregon
  - Urologic Consultants of Southeast Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Research Across America, Carrollton, Texas
  - Research Across America, Dallas, Texas
  - University of Washington, Seattle, Washington
- Germany (5):
  - University of Bonn, Clinic for Dermatology and Allergy, Bonn
  - University of Halle, Center for Reproduction and Andrology, Halle
  - Praxis Dr. Szymula, Leipzig
  - Praxis Dr. Schulze, Markkleeberg
  - University of Muenster, Center for Reproduction and Andrology, Münster

IPD SHARING:
Plan to Share IPD: No
Individual Participant data shared with associated investigational sites only.

REFERENCES:
- [Derived] Honig S, Gittelman M, Kaminetsky J, Wang C, Amory JK, Rohowsky N, Dudley RE, Woun Seo B, Newmark J, Swerdloff R. Two-Year Analysis of a New Oral Testosterone Undecanoate (TU) Formulation in Hypogonadal Men: Efficacy, Impact on Psychosexual Function, and Safety. J Sex Med. 2022 Dec;19(12):1750-1758. doi: 10.1016/j.jsxm.2022.09.002. Epub 2022 Oct 20. PMID 36272969

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Testosterone Undecanoate: Oral testosterone undecanoate 100-300 mg T BID, for 12 months.
- Transdermal Testosterone Gel (AndroGel): Transdermal testosterone gel 2.5-10 g/applied once daily for 12 months
Period: Overall Study
Arm/Group | Oral Testosterone Undecanoate | Transdermal Testosterone Gel (AndroGel)
Started | 88 | 94
Completed | 69 | 62
Not Completed | 19 | 32
Not completed — Adverse Event | 1 | 5
Not completed — Lost to Follow-up | 1 | 6
Not completed — Non-compliance with Study Drug | 3 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 4 | 12
Not completed — Hematocrit >54% | 1 | 1
Not completed — PSA increase of >1.4 ng/mL | 4 | 3
Not completed — ineligible/noncompliant/ subject reason | 4 | 4

BASELINE CHARACTERISTICS:
Population: 1. Subjects were to have completed Study CLAR-09007.
  2. Subjects were to have adequate venous access in the left or right arm to allow collection of a number of blood samples via a venous cannula.
  3. Subjects were required to remain off all forms of T except for study medication throughout the entire study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Testosterone Undecanoate | Transdermal Testosterone Gel (AndroGel) | Total
Number analyzed (Participants) | 88 | 94 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 94 | 182
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (10.04) | 56.8 (11.23) | 56.5 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 88 | 94 | 182
Region of Enrollment [Number; unit: participants]
  United States | 88 | 94 | 182

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in T Cholesterol
Description: Long-term safety profile of oral TU product compared with AndroGel based on absolute change from primary baseline based on Total Cholesterol, HDL, LDL, hemoglobin, hematocrit and prostate volume.
Time Frame: Approximately 365 days
Population: The number analyzed is less than the number of participants who began the study due to early withdrawals from study, and no available data for comparison to baseline values.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Oral TU: Subjects treated with Oral TU
- Transdermal T-gel: Subjects treated with Transdermal T-gel with a measurement taken after approximately 365 days of treatment.
Arm/Group | Oral TU | Transdermal T-gel
Number analyzed (Participants) | 68 | 62
mg/dL | 0.2 [-8.4 to 8.9] | 8.2 [-0.1 to 16.6]

2. Primary Outcome: Absolute Change From Baseline in HDL
Description: as for outcome 1
Time Frame: Approximately 365 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Oral TU | Transdermal T-gel
Number analyzed (Participants) | 68 | 62
mg/dL | 2.4 [0.7 to 4.1] | 4.0 [2.5 to 5.5]

3. Primary Outcome: Absolute Change From Baseline in LDL
Description: as for outcome 1
Time Frame: Approximately 365 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Oral TU | Transdermal T-gel
Number analyzed (Participants) | 67 | 61
mg/dL | -1.5 [-9.5 to 6.5] | 6.0 [-1.2 to 13.1]

4. Primary Outcome: Absolute Change From Baseline in Hgb
Description: as for outcome 1
Time Frame: Approximately 365 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Oral TU | Transdermal T-gel
Number analyzed (Participants) | 68 | 62
g/dL | 0.36 [0.11 to 0.61] | 0.36 [0.07 to 0.65]

5. Primary Outcome: Absolute Change From Baseline in Hct
Description: as for outcome 1
Time Frame: Approximately 365 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Oral TU | Transdermal T-gel
Number analyzed (Participants) | 68 | 62
percent | 0.38 [-0.30 to 1.06] | 0.37 [-0.44 to 1.19]

6. Primary Outcome: Absolute Change From Baseline in Prostate Volume
Description: as for outcome 1
Time Frame: Approximately 365 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cc
Arm/Group | Oral TU | Transdermal T-gel
Number analyzed (Participants) | 68 | 61
cc | 1.09 [-0.78 to 2.97] | 0.40 [-1.81 to 2.62]

ADVERSE EVENTS:
Time Frame: 365 days
Groups:
- Oral TU: Subjects treated with Oral TU with a measurement taken after approximately 365 days of treatment are used for safety laboratory values for comparisons to baseline. All subjects who received at least one dose of study drug were included in the reporting of treatment emergent adverse events.
- Transdermal T-gel: Subjects treated with Transdermal T-gel with a measurement taken after approximately 365 days of treatment are used for safety laboratory values for comparisons to baseline. All subjects who received at least one dose of study drug were included in the reporting of treatment emergent adverse events.
Arm/Group | Oral TU | Transdermal T-gel
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/94
Serious Adverse Events (participants affected / at risk) | 6/88 | 6/94
Other Adverse Events (participants affected / at risk) | 32/88 | 33/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral TU (N=88) | Transdermal T-gel (N=94)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastric ulcer hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 0 (0) | 1 (1) — Same subject as reported for prostate cancer 102-036
fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Same subject as SAE reported for Sepsis 102-036
Cerebellar Infarction (Nervous system disorders) | 1 (1) | 0 (0) — Same subject as SAE of Cerebrovascular Accident 101-043
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1) — Same subject as SAE of Cerebellar Infarction 101-043
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Alcohol detoxification (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral TU (N=88) | Transdermal T-gel (N=94)
Polycythemia (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Bronchitis (Infections and infestations) | 4 (4) | 4 (4)
Sinusitis (Infections and infestations) | 4 (4) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2)
Hematocrit Increased (Investigations) | 4 (4) | 2 (2)
PSA Increased (Investigations) | 2 (2) | 2 (2)
Hypertriglyceridemia (Investigations) | 1 (1) | 2 (2)
Arthalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Invertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days